CLINICAL TRIAL: NCT03989648
Title: Comparison of the Adequacy of Exsanguination Between Esmarch Bandages and Simple Leg Elevation in Minimally Invasive Total Knee Arthroplasty : A Randomized Controlled Trial
Brief Title: Adequacy of Exsanguination Between Esmarch Bandages and Simple Leg Elevation in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COA 028/2562
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Esmarch Bandages; Simple Leg Elevation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esmarch bandages (Active Comparator)
  Interventions: Other: Esmarch bandages
- simple leg elevation (Active Comparator)
  Interventions: Other: simple leg elevation

INTERVENTIONS:
Other: Esmarch bandages — Esmarch bandage (also known as Esmarch's bandage for surgical haemostasis or Esmarch's tourniquet) in its modern form is a narrow (5 to 10 cm wide) soft rubber bandage that is used to expel venous blood from a limb (exsanguinate) that has had its arterial supply cut off by a tourniquet.
  Arms: Esmarch bandages
Other: simple leg elevation — simple leg elevation 45 degree for 2 minutes is used to expel venous blood from a limb
  Arms: simple leg elevation

SUMMARY:
To compare the adequacy of exsanguination in the surgical field between the use of the Esmarch bandages elevation and the simple leg elevation.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee

Exclusion Criteria:

* There are deep vein thrombosis and pulmonary embolism
* There are bleeding disorder,hypercoagulability,peripheral arterial disease and chronic venous insufficiency
* Take blood clotting pills
* Have had total knee arthroplasty
* BMI > 30

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Fromme-Boezaart surgical field scale | Immediate after surgery
  Fromme-Boezaart surgical field scale is visual assessment of surgical field using a 6-point scale (min=0, max=5)
  0 mean No bleeding
  1. mean Slight bleeding ; no suctioning of blood required
  2. mean Slight bleeding ; occasional suctioning required. Surgical field not threatened
  3. mean Slight bleeding ; frequent suctioning required. Bleeding threatens surgical filed a few seconds after suction is removed
  4. mean Moderate bleeding ; frequent suctioning required. Bleeding threatens surgical field directly after suction is removed
  5. mean Severe bleeding ; constant suctioning required. Bleeding appears faster than can be removed by suction. Surgical field severely threatened and surgery not possible 0=best possible operating conditions and dryness of the surgical field; 5= worst possible conditions

SECONDARY OUTCOMES:
Numerical rating scale: NRS at 24 hrs | 24 hours after surgery
  NRS is a pain intensity assessment of patients using a 11 point scale (min=0, max=10) 0=no pain 10= worst pain
Numerical rating scale: NRS at 72 hrs | 72 hours after surgery
  NRS is a pain intensity assessment of patients using a 11 point scale (min=0, max=10) 0=no pain 10= worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand

REFERENCES:
- [Derived] Chaitantipongse S, Hongku N, Thiengwittayaporn S. Optimizing surgical field visualization in total knee arthroplasty: a randomized controlled trial comparing esmarch bandages and simple leg elevation. J Orthop Surg Res. 2025 May 13;20(1):455. doi: 10.1186/s13018-025-05853-6. PMID 40355975